CLINICAL TRIAL: NCT05067816
Title: Scaling up the Med-South Lifestyle Program to Reduce Chronic Disease in Partnership With Rural Communities: Phase 2
Brief Title: Med-South Lifestyle Program Implementation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-1281
Record Dates: First submitted 2021-09-23; First posted 2021-10-05 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-09

CONDITIONS: Healthy Lifestyle

STUDY DESIGN:
Intervention Model Description: Effectiveness-implementation hybrid Type 3 study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Distance Scale-Up Format (Active Comparator): 10 sites with up to 150 program participants will be randomly assigned to a distance scale-up format where each site implementation team will receive technical assistance individually. All implementation training will occur using a virtual web-based format. Implementation teams will receive 8 hours of web-conferences, 2 hours of online training, and 4 hours of technical assistance.
  Interventions: Behavioral: Med-South Lifestyle Program
- Quality Improvement Collaborative Scale-Up Format (Experimental): 10 sites with up to 150 program participants will be randomly assigned to a quality improvement collaborative scale-up format where implementation teams will work collaboratively during training and implementation. All implementation training will occur using a virtual web-based format. Implementation teams will receive 8 hours of web-conferences, 2 hours of online training, and 4 hours of technical assistance.
  Interventions: Behavioral: Med-South Lifestyle Program

INTERVENTIONS:
Behavioral: Med-South Lifestyle Program — The Med-South Lifestyle Program (MSLP) is an evidence-based behavior change intervention that translates the PREDIMED (Mediterranean) dietary pattern for a southeastern US population and includes support for increased physical activity. To promote healthy dietary intake and increased physical activity, the intervention incorporates theory-based behavioral approaches targeting self-efficacy, self-regulation, and internal motivation. The MSLP is delivered in 4 monthly counseling sessions with 3 interim phone follow-up contacts. A maintenance phase lasting 6 months follows the 4-month MSLP and includes 2 phone contacts about 2 months apart. Participants are counseled individually, with 2 in-person counseling visits (at the 1st and 4th counseling visit) and 5 total phone contacts. Each participant is provided with program materials in a participant manual, a cookbook, and a local resource manual identifying community resources to support making targeted behavior changes.
  Other Names: Med-South Program

SUMMARY:
The purpose of this study is to determine the processes by which a previously proven lifestyle intervention (the Med-South Lifestyle Program) can most effectively and efficiently be translated into public health and clinical practice to positively impact chronic disease risk reduction among mostly minority, rural, and medically underserved populations.

DETAILED DESCRIPTION:
Purpose: Although lifestyle behavior change interventions are widely recommended to improve health, they are not being implemented sufficiently or equitably on a national scale, particularly in rural communities. The research team has developed and tested multiple lifestyle interventions, which have culminated in the Med-South Lifestyle Program (MSLP), an evidence-based behavior change intervention that translates the Prevention with Mediterranean Diet (PREDIMED) dietary pattern for a Southeastern US population and includes support for increased physical activity. In this research, the investigators propose to identify the most effective and efficient way to scale-up the MSLP for use in public health and clinical practices settings so that it reaches minority, rural, and medically underserved populations. In Phase 2, the investigators will apply an effectiveness-implementation hybrid design to compare two formats for scaling up MSLP on implementation outcomes (primary aim) and confirm the MSLP's impact on behavioral and clinical outcomes (secondary aim).

Participants: Phase II participants include: staff at 20 rural North Carolina sites (10 health departments and 10 federally qualified health centers) and participants from each site (15 each, 300 total)

Procedures (methods): Test the effects of scaling up MSLP using two different formats. Using an effectiveness-implementation hybrid Type 3 design, the investigators will randomize 20 sites (10 health departments and 10 Federally Qualified Health Centers (FQHCs)) to 1 of 2 formats for delivering scale up strategies: distance (webinar and phone) vs. a blended in-person/distance collaborative format. Each site will collect data on 15 patients (n=300).

Aim 1: Site level: compare the relative effects of the 2 scale-up formats on implementation outcomes (reach, acceptability, feasibility, fidelity, and cost).

Aim 2: Participant-level: assess changes in behavioral and clinical outcomes: (1) self-reported diet and physical activity and (2) weight from baseline to follow-up (4 and 10 months). Compare outcomes across the 2 scale-up delivery formats.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* English speaking (Spanish-speaking only in selected sites with bilingual staff)
* Ages 18-80

Exclusion Criteria:

* Malignancy
* Advanced kidney disease (estimated creatinine clearance < 30 mL/min)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Percentage of Eligible Patients Participating | Month 10
  Percentage of each setting's eligible patients who participate in the Med-South Lifestyle Program and the representativeness of participants (age, gender, race/ethnicity) as compared to overall population of eligible patients.
Percentage of Med-South Lifestyle Program Delivered as Intended | Month 10
  To determine delivery fidelity, the study team will measure the degree to which the intervention is delivered as intended as assessed by direct observations and audio file reviews documented by checklist.

SECONDARY OUTCOMES:
Mean Change in Number of Fruit and Vegetable Servings Per Day | Month 0, Month 10
  The mean difference in fruit and vegetable servings per day (baseline servings/day - follow-up servings/day) as measured by the Block Fruit-Vegetable-Fiber Screener.
  The Block Fruit-Vegetable-Fiber Screener is a 10-item scale with responses ranging from: (1) Less than 1/week to (5) 2+ a day. Higher scores reflect a better outcome.
Mean Change in Minutes of Physical Activity Per Week | Month 0, Month 10
  Mean difference in minutes of physical activity per week (baseline activity in minutes/week - follow-up activity in minutes/week) as measured by the validated modified RESIDE questionnaire. The RESIDE questionnaire is a 21-item self-administered instrument in which participants recall the frequency, duration, and destination of their walking (for transport and recreation) within and outside of their neighborhood, and cycling activity in a usual week. Higher scores indicate more minutes of activity.
Mean Percent Change in Weight | Month 0, Month 10
  Mean weight change (in kg) from baseline to follow-up expressed as a percentage of baseline weight
Mean Change in Systolic Blood Pressure at end of 4-Month Med-South Program | Month 0, Month 4
  Mean difference in systolic blood pressure measured at session 1 and at the end of the Med-south Program (session 4).
Mean Change in Systolic Blood Pressure at end of 6-Month Maintenance Phase | Month 4, Month 10
  Mean difference in systolic blood pressure measured at session 4 of the Med-South Program and at the end of the maintenance phase (month 10).
Mean Change in Diastolic Blood Pressure at end of 4-Month Med-South Program | Month 0, Month 4
  Mean difference in diastolic blood pressure measured at session 1 and at the end of the Med-South Program (session 4).
Mean Change in Diastolic Blood Pressure at end of 6-Month Maintenance Phase | Month 4, Month 10
  Mean difference in diastolic blood pressure measured at session 4 of the Med-South Program and at the end of the maintenance phase (month 10).

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Samuel-Hodge, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Jennifer Leeman, DrPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina at Chapel Hill (UNC).
Supporting Information: Study Protocol, SAP
Time Frame: 9 to 36 months following publication
Access Criteria: Investigator who proposes to use the data must have approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and execute a data use/sharing agreement with UNC.
URL: http://research.unc.edu/clinical-trials/clinical-trials-gov/icmje/

REFERENCES:
- [Background] Samuel-Hodge CD, Gizlice Z, Allgood SD, Bunton AJ, Erskine A, Leeman J, Cykert S. Strengthening community-clinical linkages to reduce cardiovascular disease risk in rural NC: feasibility phase of the CHANGE study. BMC Public Health. 2020 Feb 21;20(1):264. doi: 10.1186/s12889-020-8223-x. PMID 32085707
- [Background] Leeman J, Calancie L, Hartman MA, Escoffery CT, Herrmann AK, Tague LE, Moore AA, Wilson KM, Schreiner M, Samuel-Hodge C. What strategies are used to build practitioners' capacity to implement community-based interventions and are they effective?: a systematic review. Implement Sci. 2015 May 29;10:80. doi: 10.1186/s13012-015-0272-7. PMID 26018220
- [Background] Keyserling TC, Samuel-Hodge CD, Pitts SJ, Garcia BA, Johnston LF, Gizlice Z, Miller CL, Braxton DF, Evenson KR, Smith JC, Davis GB, Quenum EL, Elliott NT, Gross MD, Donahue KE, Halladay JR, Ammerman AS. A community-based lifestyle and weight loss intervention promoting a Mediterranean-style diet pattern evaluated in the stroke belt of North Carolina: the Heart Healthy Lenoir Project. BMC Public Health. 2016 Aug 5;16:732. doi: 10.1186/s12889-016-3370-9. PMID 27495295
- [Background] Cubillos L, Estrada Del Campo Y, Harbi K, Keyserling T, Samuel-Hodge C, Reuland DS. Feasibility and Acceptability of a Clinic-based Mediterranean-style Diet Intervention to Reduce Cardiovascular Risk for Hispanic Americans With Type 2 Diabetes. Diabetes Educ. 2017 Jun;43(3):286-296. doi: 10.1177/0145721717706030. Epub 2017 Apr 21. PMID 28427311
- [Background] Thomas T, Samuel-Hodge CD, Porterfield DS, Alva ML, Leeman J. Scaling Up Diabetes Prevention Programs in North Carolina: Perceptions of Demand From Potential Program Recipients and Providers. Diabetes Educ. 2019 Feb;45(1):116-124. doi: 10.1177/0145721718811564. Epub 2018 Nov 9. No abstract available. PMID 30413136
- [Background] Rohweder C, Wangen M, Black M, Dolinger H, Wolf M, O'Reilly C, Brandt H, Leeman J. Understanding quality improvement collaboratives through an implementation science lens. Prev Med. 2019 Dec;129S:105859. doi: 10.1016/j.ypmed.2019.105859. Epub 2019 Oct 23. PMID 31655174
- [Background] Leeman J, Toles M. What does it take to scale-up a complex intervention? Lessons learned from the Connect-Home transitional care intervention. J Adv Nurs. 2020 Jan;76(1):387-397. doi: 10.1111/jan.14239. Epub 2019 Nov 20. PMID 31642091
- [Derived] Samuel-Hodge CD, Pham L, Lyons K, Draeger LB, Jiang L, Lin FC, Ram R, Leeman J. Scaling up the Med-South Lifestyle Program in public health settings to reduce chronic disease risk: a hybrid implementation-effectiveness study. Front Public Health. 2025 Jun 5;13:1564567. doi: 10.3389/fpubh.2025.1564567. eCollection 2025. PMID 40538692
- See also: The current study will adapt intervention and dissemination materials from the CHANGE Study. — http://change.web.unc.edu/

DOCUMENTS (1):
  • Informed Consent Form (2021-07-27): https://cdn.clinicaltrials.gov/large-docs/16/NCT05067816/ICF_000.pdf